CLINICAL TRIAL: NCT01404494
Title: Testing Subjects With Traumatic Brain Injury Using Haptic Technology
Brief Title: Testing Devices That Involve the Sense of Touch in Subjects With Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 110137; 11-CC-0137
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2015-02-06

CONDITIONS: Traumatic Brain Injury
Keywords: Haptic Skills; Computer Assisted Interface; TBI; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Previous studies have shown that computer-based devices that simulate everyday tasks can be helpful for evaluation and rehabilitation in people who have had strokes. Researchers are interested in studying whether similar devices can be used to evaluate and treat individuals who have had a traumatic brain injury, to determine if the device should be developed to help with rehabilitation in the future.

Objectives:

- To evaluate the effectiveness of a computer-based simulation compared with actual performance of actions in individuals who have had a traumatic brain injury.

Eligibility:

- Individuals at least 18 years of age who have had a non-penetrating mild or moderate traumatic head injury within the past year and have experience playing computer games.

Design:

* Participants will be screened with a physical and neurological examination and medical history.
* Participants will complete questionnaires and an interview about mood and feelings, stress levels, quality of life, and how well they function at work or at home. Participants will also have tests of memory, attention, thinking, and reasoning. Some of the questionnaires and tests will be completed in writing, some orally, and some on a computer.
* Participants will have movement and coordination tests that involve simple tasks such as putting pegs in a pegboard, using a key, lifting different objects, and folding things.
* Participants will duplicate the movement and coordination tests by using a computer program that simulates the tasks with a cursor on a computer screen. Participants will do four separate simulated tasks (such as arranging letters or hitting a nail with a hammer) three times.
* The full visit will take about 4 hours, and no followup visits are required.

DETAILED DESCRIPTION:
Adults who have suffered traumatic brain injury are people who have a wide variety of signs and symptoms. These often include problems with motor planning and learning, memory, cognitive performance and behavior. The physical findings and self reports of symptoms are heterogeneous, and do not always correlate with anatomic findings. Evaluation and measurement of function in this population, and treatment of functional deficits are being developed so that treatments can be specifically targeted toward functional recovery. Additionally, evaluation and treatment usually relies heavily on labor intensive interventions. This study will assess the feasibility of using haptic devices that interface the user via touch using force as feedback in subjects with a TBI. Haptic devices are similar to joysticks. The specific haptic device we are using in this project is a stylus, shaped like a pen with which the subject navigates virtual space moving a cursor on a computer screen. The project aims to obtain pilot data in relation to how an individual with TBI performs measuring their engagement and interaction with the haptic, which is programmed to simulate functional activity and cognitive tasks, and whether the haptic devices can reliably be used for data capture.

Study Population

Seventy adult subjects with a clinical diagnosis of a non-penetrating TBI will be enrolled. Subjects will need to be at least 1 year from date of initial brain injury. Subjects will be recruited from NIH, affiliated hospitals/clinics, and in the community.

Design

This is a prospective cohort study of subjects with a clinical diagnosis of a non-penetrating traumatic brain injury. Subjects will be recruited and assessed at the National Institutes of Health. Data will be shared and stored at NIH. Subjects will be stratified according to findings into cohorts for comparison. Subjects will not be treated with experimental therapies as part of the research study.

The role of multimodal visuo-sensory motor input learning using haptic devices will be explored in this project. Virtual reality has been applied to both the evaluation and treatment of persons with TBI. The application of simulated environments has helped engage patients in therapeutic activities and also has provided real life situations that call for integration of sensory, cognitive and motor activities Haptic and robotic devices, which provide sensory and force input to assist in human movement, have been used to help in neurorecovery.

Each subject will have only one test session and there will be no further follow-up appointments. The haptic session is designed to take no more than 1 hour. However, it may take longer for some to complete the battery of tests. It may take up to four hours to complete the NIH processes such as admissions, the history and physical, and the haptic session.

Outcome Measures

Performance on haptic tasks will be assessed for time to completion, distance of trajectories and frequency of repeated trajectories.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects eligible for participation in this research study must meet the following inclusion criteria:

Ages 18 and older

Some experience with computer games

Diagnosis of traumatic brain injury

At least 1 year from initial traumatic brain injury

Able to understand and comply with study procedures

Able to read, speak, and understand English

Capable of providing own consent

EXCLUSION CRITERIA:

Subjects are not eligible for participation in this research study if any of the following conditions exist:

Inability to grasp and manipulate a 2 cm diameter pen like structure with preferred hand

Unable to adequately detect objects on the computer screen

Penetrating head injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04-05; Study Completion 2015-02-06

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aisen ML, Krebs HI, Hogan N, McDowell F, Volpe BT. The effect of robot-assisted therapy and rehabilitative training on motor recovery following stroke. Arch Neurol. 1997 Apr;54(4):443-6. doi: 10.1001/archneur.1997.00550160075019. PMID 9109746
- [Background] Broeren J, Rydmark M, Sunnerhagen KS. Virtual reality and haptics as a training device for movement rehabilitation after stroke: a single-case study. Arch Phys Med Rehabil. 2004 Aug;85(8):1247-50. doi: 10.1016/j.apmr.2003.09.020. PMID 15295748
- [Background] Broeren J, Sunnerhagen KS, Rydmark M. A kinematic analysis of a haptic handheld stylus in a virtual environment: a study in healthy subjects. J Neuroeng Rehabil. 2007 May 9;4:13. doi: 10.1186/1743-0003-4-13. PMID 17490470